CLINICAL TRIAL: NCT00672737
Title: Experimental Pain Processing and Autonomic Function in Subjects Suffering From Obstructive Sleep Apnea
Brief Title: Study of Pain Processing in Subjects Suffering From Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anthony Doufas, MD, PhD, Stanford University
Other Study IDs: SU-01222008-985; 10374
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-01

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Remifentanil; Drug Tolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Males at risk for OSA: Males at risk for obstructive sleep apnea were invited to have a "sleep study" either at home or at Stanford Sleep Center.
  A week after their sleep study (Polysomnography), all volunteers underwent quantitative sensory testing in the laboratory, during which their pain thresholds and tolerances to heat (Heat pain threshold and tolerance) and cold (Cold pain threshold and tolerance) stimuli were assessed, under two different concentrations (1 and 2 mcg/mL, in randomized order) of remifentanil, a short-acting opioid, given as a computer-controlled infusion.
  Interventions: Drug: Remifentanil; Procedure: Cold pain threshold and tolerance; Device: Heat pain threshold and tolerance; Procedure: Polysomnography

INTERVENTIONS:
Drug: Remifentanil — Remifentanil was administered as a computer-controlled infusion, targeting two different effect site concentrations, 1 and 2 mcg/mL, in randomized order.
Procedure: Cold pain threshold and tolerance — Ice water was used to assess cold-related pain threshold and tolerance, defined as the time that the volunteers could keep their hands in the water before they started feeling pain or this feeling becomes unbearable, for threshold and tolerance, respectively.
Device: Heat pain threshold and tolerance — TSAII Neuroanalyzer (Medoc Advanced Medical Systems, Durham, NC), was used to assess the heat-related pain and tolerance of the volunteers defined as the respective temperatures where they started feeling as painful or unbearable.
Procedure: Polysomnography — All volunteers underwent a polysomnography study at home or at Stanford Sleep Center, approximately one week before their experimental pain assessment in the laboratory
  Other Names: sleep study

SUMMARY:
We would like to test the effect of opioid medication on pain sensitivity in subjects who have been diagnosed with a sleep disorder called Obstructive Sleep Apnea (OSA) compared to other subjects without OSA. Patients with OSA may have an altered sensitivity to the sedative, analgesic, and respiratory depressant effects of opioids.

DETAILED DESCRIPTION:
The purpose of the study is to test the hypothesis that patients who suffer from moderate-to-severe OSA have increased pain thresholds and are more sensitive to the analgesic effects of opioids compared to patients with normal sleep-related breathing physiology. We will evaluate the effect of remifentanil, a short acting mu-opioid receptor agonist, on pain using an experimental heat and cold-induced pain tests, and compare it between volunteers with and without a polysomnography (PSG)-based diagnosis of obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:1. Male 2 .18 - 55 years of age 3. Body mass index (BMI) lower or equal to 30 kg/m2 4. Absence of severe systemic disease that results in functional limitations (i.e. poorly controlled hypertension, angina pectoris, prior myocardial infarction, pulmonary disease that limits activity) 5.Subjects must be able to comprehend spoken and written English

Exclusion Criteria:1. Major psychiatric, neurological, or neuromuscular disorder 2. Known diabetes mellitus or thyroid disease 3. Allergy to study medication (remifentanil) 4. History of addiction 5. Alcohol consumption which exceeds 2 drinks per day and /or drug abuse. 6. Chronic or acute use of opioids, or other medications affecting the CNS.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Males at risk for obstructive sleep apnea (OSA). We invited male volunteers (18 55 years old) with a history of habitual snoring and/or a formal diagnosis of OSA to participate in a study evaluating sleep and experimental pain processing.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Doufas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Doufas AG, Tian L, Padrez KA, Suwanprathes P, Cardell JA, Maecker HT, Panousis P. Experimental pain and opioid analgesia in volunteers at high risk for obstructive sleep apnea. PLoS One. 2013;8(1):e54807. doi: 10.1371/journal.pone.0054807. Epub 2013 Jan 29. PMID 23382975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2008 till March 2010, we invited male volunteers (18-55 years old) with a history of habitual snoring and/or a formal diagnosis of OSA to participate in a study evaluating sleep and experimental pain processing at the Human Pain Laboratory in the Department of Anesthesiology at Stanford University.
Pre-assignment Details: We screened 167 male volunteers; 56 consented to participate to the study.
Groups:
- Male Volunteers at Risk for Sleep Apnea: After approval from the Institutional Review Board and informed consent, we assessed cold and heat pain thresholds in volunteers after overnight polysomnography (PSG). We measured insulin growth factor binding protein-1 (IGFBP-1) a hypoxia-related serum marker. Pain tests were performed at baseline, placebo, and two effect site concentrations of remifentanil (1 and 2 mg/ml), an mu-opioid agonist. Linear mixed effects regression model was employed to evaluate the association of the lowest oxyhemoglobin saturation (SaO2) during sleep and IGFBP-1 with the changes in pain thresholds after remifentanil administration.
Period: Overall Study
Arm/Group | Male Volunteers at Risk for Sleep Apnea
Started | 56
Completed | 48
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: 56 volunteers signed informed consent; 3 of withdrew before participation in any procedure. The remaining 53 who underwent a polysomnography study are included for Baseline Characteristics.
Arm/Group | Male Volunteers at Risk for Sleep Apnea
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 53
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 53
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Experimental Cold-induced Pain - IGFBP-1
Description: The effect of insulin growth factor binding protein-1 (IGFBP-1), a serum hypoxia marker, on the change of cold-induced pain thresholds under remifentanil was estimated using a mixed linear regression model. The results were expressed by the estimated beta (95% CI), indicating how much the change in the cold pain threshold (expressed in seconds) under remifentanil, was altered per unit of change in the IGFBP-1. For example, for every 1-pg/mL increase in the serum level of IGFBP-1, cold pain threshold will additionally increase by 0.0025 seconds for every 1-mcg/mL increase in the plasma level of remifentanil.
Time Frame: 2 to 3 weeks
Population: Volunteers with evaluable data were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: [sec/(mcg/mL)] /pg/mL
Groups:
- at Risk for Sleep Apnea: After approval from the Institutional Review Board and informed consent, we assessed cold and heat pain thresholds in volunteers after overnight polysomnography (PSG). We measured insulin growth factor binding protein-1 (IGFBP-1) a hypoxia-related serum marker. Pain tests were performed at baseline, placebo, and two effect site concentrations of remifentanil (1 and 2 mg/ml), an mu-opioid agonist. Linear mixed effects regression model was employed to evaluate the association of the lowest oxyhemoglobin saturation (SaO2) during sleep and IGFBP-1 with the changes in pain thresholds after remifentanil administration.
Arm/Group | at Risk for Sleep Apnea
Number analyzed (Participants) | 48
[sec/(mcg/mL)] /pg/mL | 0.0025 [0.0009 to 0.0041]
Statistical Analysis 1: Comparison: at Risk for Sleep Apnea; Beta for IGFBP-1: for every 1-pg/mL increase in its serum level the cold pain threshold will additionally increase by 0.0025 seconds for every 1-mcg/mL increase in the plasma level of remifentanil; Test type: Superiority or Other; p < 0.05, Regression, Linear; Adjusted for body mass index, age of the volunteers, and a binary variable indicating the type (home-based vs. in-laboratory); Slope = 0.0025, 95% CI 2-sided [0.0009 to 0.0041] — Mixed linear regression
Statistical Analysis 2: Comparison: at Risk for Sleep Apnea; Beta for SaO2: for every 1-%-absolute decrease in the nadir SaO2 the cold pain threshold will additionally increase by 0.9694 seconds for every 1-mcg/mL increase in the plasma level of remifentanil; Test type: Superiority or Other; p = 0.05, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Slope = -0.9694, 95% CI 2-sided [-1.9127 to -0.0261] — Mixed linear regression

2. Primary Outcome: Experimental Heat-induced Pain - IGFBP-1
Description: The effect of arterial oxyhemoglobin desaturation during sleep (chronic intermittent hypoxia expressed by insulin growth factor binding protein-1 (IGFBP-1), a serum hypoxia marker, on the change of heat-induced pain thresholds under remifentanil was estimated using a mixed linear regression model. The results were expressed by the estimated betas (95% CI), indicating how much the change in the heat pain threshold (expressed in C') under remifentanil, was altered per unit of change in the IGFBP-1. For example, for every 1-pg/mL increase in serum level of IGFBP-1, the heat pain threshold will additionally decrease by 0.0001 'C for every 1-mcg/mL increase in the plasma level of remifentanil.
Time Frame: 2 to 3 weeks
Population: Volunteers with evaluable data were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: ['C/(mcg/mL)] /pg/mL
Groups:
- Males at Risk for OSA: Males at risk for obstructive sleep apnea were invited to have a "sleep study" either at home or at Stanford Sleep Center.
  A week after their sleep study (Polysomnography), all volunteers underwent quantitative sensory testing in the laboratory, during which their pain thresholds and tolerances to heat (Heat pain threshold and tolerance) and cold (Cold pain threshold and tolerance) stimuli were assessed, under two different concentrations (1 and 2 mcg/mL, in randomized order) of remifentanil, a short-acting opioid, given as a computer-controlled infusion.
  Remifentanil: Remifentanil was administered as a computer-controlled infusion, targeting two different effect site concentrations, 1 and 2 mcg/mL, in randomized order.
Arm/Group | Males at Risk for OSA
Number analyzed (Participants) | 48
['C/(mcg/mL)] /pg/mL | -0.0001 [-0.0001 to -0.0001]
Statistical Analysis 1: Comparison: Males at Risk for OSA; Beta for IGFBP-1: for every 1-pg/mL increase in its serum level, the heat pain threshold will additionally decrease by 0.0001 'C for every 1-mcg/mL increase in the plasma level of remifentanil; Test type: Superiority or Other; p < 0.05, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Slope = -0.0001, 95% CI 2-sided [-0.0001 to -0.0001] — Mixed linear regression
Statistical Analysis 2: Comparison: Males at Risk for OSA; Beta for SaO2: for every 1-%-absolute decrease in the nadir SaO2, the heat pain threshold will additionally increase by 0.0172 'C for every 1-mcg/mL increase in the plasma level of remifentanil; Test type: Superiority or Other; p < 0.05, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Slope = -0.0172, 95% CI 2-sided [-0.018 to 0.0556] — Mixed linear regression

3. Primary Outcome: Experimental Cold-induced Pain - SaO2
Description: The effect of arterial oxyhemoglobin desaturation during sleep (chronic intermittent hypoxia expressed by nadir SaO2 during polysomnography) on the change of cold-induced pain thresholds under remifentanil was estimated using a mixed linear regression model. The results were expressed by the estimated betas (95% CI), indicating how much the change in the cold pain threshold (expressed in seconds) under remifentanil, was altered per unit of change in the SaO2. For example, for every 1-%-absolute decrease in the nadir SaO2, the cold pain threshold will additionally increase by 0.9694 seconds for every 1-mcg/mL increase in the plasma level of remifentanil.
Time Frame: 2 to 3 weeks
Population: Volunteers with evaluable data were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: [sec/(mcg/mL)] /%
Arm/Group | at Risk for Sleep Apnea
Number analyzed (Participants) | 48
[sec/(mcg/mL)] /% | -0.9694 [-1.9127 to -0.0261]

4. Primary Outcome: Experimental Heat-induced Pain - SaO2
Description: The effect of arterial oxyhemoglobin desaturation during sleep (chronic intermittent hypoxia expressed by nadir SaO2 during polysomnography), on the change of heat-induced pain thresholds under remifentanil was estimated using a mixed linear regression model. The results were expressed by the estimated betas (95% CI), indicating how much the change in the heat pain threshold (expressed in C') under remifentanil, was altered per unit of change in the SaO2. For example, for every 1-%-absolute decrease in the nadir SaO2, the heat pain threshold will additionally increase by 0.0172 'C for every 1-mcg/mL increase in the plasma level of remifentanil.
Time Frame: 2 to 3 weeks
Population: Volunteers with evaluable data were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: ['C/(mcg/mL)] /%
Arm/Group | Males at Risk for OSA
Number analyzed (Participants) | 48
['C/(mcg/mL)] /% | -0.0172 [-0.018 to 0.0556]

ADVERSE EVENTS:
Arm/Group | at Risk for Sleep Apnea
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes